CLINICAL TRIAL: NCT01533480
Title: A Prospective, Double-masked, Placebo Controlled Comparison of Topical 0.15% Ganciclovir Gel (Zirgan®) Versus 0.3% Hypromellose Gel (Genteal Gel®; Placebo) for the Treatment of Adenovirus Conjunctivitis
Brief Title: A Placebo Controlled Comparison of Topical Zirgan Versus Genteal Gel for the Treatment of Adenovirus Conjunctivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lifelong Vision Foundation (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADV-GAN-10-2011; pro00006720 (Registry Identifier: Chesapeake IRB)
Record Dates: First submitted 2012-01-31; First posted 2012-02-15 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Keratoconjunctivitis Due to Adenovirus; Viral Shedding
Keywords: Adenovirus; Conjunctivitis; keratoconjunctivitis; viral shedding; subepithelial infiltrate; bulbar injection
MeSH Terms: conditions — Adenoviridae Infections; Conjunctivitis; Keratoconjunctivitis | interventions — Ganciclovir; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zirgan, Adenovirus conjunctivitis, (Active Comparator): Zirgan
  Interventions: Drug: Zirgan
- genteal gel (Placebo Comparator): 0.3% Hypromellose gel (genteal gel)
  Interventions: Drug: genteal gel

INTERVENTIONS:
Drug: Zirgan — 0.15% ganciclovir gel(Zirgan)
  Other Names: Virgan
  Arms: Zirgan, Adenovirus conjunctivitis,
Drug: genteal gel — 0.3% Hypromellose gel
  Other Names: genteal
  Arms: genteal gel

SUMMARY:
The investigators are conducting this study because the patient have an eye infection which is called adenoviral conjunctivitis, and is the most common cause of "pink eye". There is currently no treatment for this condition. However, the researchers associated with this study want to understand if using a product called Zirgan, which is a topical ointment that is already FDA-approved for other types of eye infections, will help with the type of infection that the patient currently have. Zirgan is not FDA-approved to treat your type of eye infection. Your participation in this study is expected to last 21 days but the patient will only apply the topical ointment for 14 of those days. During the study, the patient will be asked to come into this clinic 8 times.

The purpose of this study is to determine whether topical Zirgan can reduce days that the patient suffers from the eye infection, and also to see if it can prevent the infection from spreading to your second eye and to also see if it can prevent the spreading of the infection to people that the patient come in close contact with.

Zirgan will be compared to Genteal Gel in this trial. Genteal Gel is a non-prescription eye lubricant gel and is commonly used for treatment of dry eye.

The patient will be asked to apply a topical ointment (either Zirgan or Genteal gel 5 times a day for the first 7 days and then 3 times a day for the following 7 days. The patient will be asked to return to the clinic 21 days after the patient starts the study for a final check-up.

It is planned that about 80 people with Adenovirus Conjunctivitis will be enrolled in this study between 8-12 sites across the United States.

The patient will be assigned to either Zirgan or Genteal gel by chance which is similar to flipping a coin.

The study groups will be assigned in a 1:1 ratio. Neither the patient nor the study doctor or study staff will be able to pick which study group The patient is in. The patient will not know and the study doctor or study staff will not know which study group the patient is in. The study doctor or study staff can find out if it is necessary to know for your health. If this happens, the study doctor or study staff may not be able to tell the patient which study group the patient was in until everyone finishes the study.

DETAILED DESCRIPTION:
Study Objectives To evaluate the safety and efficacy of 0.15% ganciclovir gel (Zirgan®) in patients with adenoviral keratoconjunctivitis in comparison with 0.3% hypromellose gel (Genteal gel®) as placebo.

Background Adenoviruses are the most common cause of ocular viral infection worldwide. Conjunctivitis and keratoconjunctivitis caused by adenoviruses are highly contagious. Adenovirus is a non-enveloped, double-stranded DNA virus comprised of 53 serotypes. Unlike many enveloped viruses which can be more easily inactivated, adenoviruses are resilient to disinfection and are long lasting on fomites. The ocular infection generally begins unilaterally and, in many cases, spreads to both eyes. It may cause epidemics and endemics, being most commonly spread in the summer or winter. Epidemics are common in day care centers, schools and the military and have been spread in the offices of eye care professionals. Patients may have painful conjunctival membranes and palpable preauricular adenopathy. Subsequent subepithelial corneal infiltrates can cause light sensitivity, reduced vision and lead to irregular astigmatism. The differential diagnosis includes herpes simplex, Chlamydia and enteroviral infection.

There are 3 major presentations of ocular adenovirus infection: Follicular conjunctivitis (predominantly serotypes 3, 4,7a); epidemic keratoconjunctivitis (EKC; predominantly serotypes 8, 19, 37, 53); and pharyngealconjunctival fever (mostly serotypes 3, 4, 7a, 11).

There is supporting laboratory and clinical data to warrant a clinical trial of topical ganciclovir for the treatment of adenoviral keratoconjunctivitis. Several studies has shown that ganciclovir (GCV) is active in vitro against adenovirus.

Primary Outcome The primary outcome of the study is to determine whether topical 0.15% ganciclovir (Zirgan®) gel alone will reduce the duration of viral shedding from the ocular surface, as determined by quantitative viral isolation in A549 cell tissue culture, compared to placebo 0.3% hypromellose gel (Genteal gel®).

Secondary Outcomes The secondary outcomes of the study are whether topical 0.15% ganciclovir will (1) reduce the incidence and severity of second eye involvement, (2) reduce the incidence and severity of subepithelial infiltrates, (3) reduce the secondary spread to family members, friends, classmates or co-workers (The virus is very stable at room temperature and can last for days on fomites, like towels, doorknobs, etc), (4) reduce the degree of bulbar conjunctival injection (redness of the eye, as determined by the Efron scale in the Appendix 2), (5) reduce ocular discomfort, and (6) be considered an effective treatment by the patient.

Sample Size The sample size for this study is based on the objective to demonstrate a statistically significant difference in the primary outcome measure (i.e., time to viral eradication). Approximately 350 subjects will be screened with Rapid Pathogens Screening (RPS) Adeno Detector Plus Immunoassay for adenovirus (applied to the conjunctiva of the most involved eye) to allow recruitment of approximately 80 RPS positive subjects in this study, with approximately 40 subjects per treatment group (randomization ratio of 1:1), in anticipation of approximately 40 culture positive subjects per treatment group (assuming a 100% culture positivity rate) and 38 of these culture positive subjects per treatment group completing the study (assuming a 5% dropout rate).

Thirty eight viral positive culture subjects per treatment group yields 90% power to detect a statistically significant difference in time of viral eradication between ganciclovir gel 0.15% and placebo (hypromellose gel) assuming: (1) a mean time to viral eradication of 7.0 days in the placebo group and 5.5 days in the ganciclovir group, (2) an estimated standard deviation of 2.0 days for both groups, and (3) using a two-sided α = 0.05 (two sample comparison of means).

The estimate of approximately 320 to 350 screenings to find approximately 80 RPS positive subjects was based on previous studies documenting approximately 25% prevalence of adenoviral conjunctivitis among patients with acute conjunctivitis. The estimated mean time to viral eradication of 7.0 days for the placebo was based on a placebo arm of a previous study evaluating the safety and efficacy of cidofovir in the treatment of viral epidemic keratoconjunctivitis and the estimated mean time to viral eradication of 5.5 days was based on assumed clinically significant decrease of 1.5 days compared to the placebo arm.

Virological Studies At the first study visit, the lower palpebral conjunctiva of each eye will be rubbed six to eight times using the Rapid Pathogen Screening (RPS) Adeno Detector Plus Immunoassay device. A positive result in the most involved eye is required to meet entry criteria. For patients entered and randomized into the treatment or placebo arms, further virologic studies for quantitative culture, PCR confirmation and viral serotyping using DNA sequencing will be performed,

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 14 years of age or older. Patients under age 18 will require parental consent for entry.
2. Give written informed consent and use or release of health and research study information.
3. Patients must be able and willing to comply with all treatment and follow-up/study procedures.
4. Patients must have a follicular conjunctivitis and present within 3 days of the onset of symptoms in the first eye.
5. Patients must agree not to wear contact lenses for 14 days while taking study medications.

Exclusion Criteria:

1. Severe dry eye or Sjögren's Syndrome.
2. Corneal graft in either eye.
3. Participation in an investigational study within the past 30 days.
4. Inability to understand instructions or comply with the study visit schedule.
5. Uniocular vision status.
6. Best corrected visual acuity worse than 20/200 in either eye.
7. Uveitis or iritis which requires treatment with corticosteroids.
8. Mucopurulent discharge.
9. Signs of any other viral, fungal, bacterial infection.
10. Congenital, acquired, or iatrogenic immune deficiency.
11. Treatment with systemic or topical ocular antiviral agents or systemic or topical steroids or topical ocular NSAIDS during the prior 14-day period.
12. Presence of subepithelial infiltrates.
13. Bilateral eye involvement with a bulbar conjunctival score of moderate or severe in both the eyes. (Grade 3 or 4 as scored using Efron scale of the bulbar hyperemia component of conjunctivitis).
14. Pregnancy test positive for women of child bearing age or women breastfeeding children or women not practicing accepted method(s) of contraception.
15. Active allergic conjunctivitis
16. History of atopic disease.
17. Known hypersensitivity or allergy to ganciclovir or to BAK or to any of the ingredients in the study drugs
18. Acute eye trauma.
19. Contact lens only with no spectacles available.
20. Expected to require concurrent ocular therapy with immunosuppressants (e.g., Restasis) during the study or have used ocular immunosuppressants within 30 days prior to study start.
21. Ocular surgery (including laser surgery) in either eye within six weeks prior to entry into this study.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Time to Viral Eradication | 14 days
  Time to viral eradication from the ocular surface, as determined by quantitative viral isolation in A549 cell tissue culture (performed on Day 0, 2, 4, 6, 8, 10, and 14)

SECONDARY OUTCOMES:
Development of sub-epithelial infiltrates | 21 days
  Development of sub-epithelial infiltrates (SEIs)-incidence for the study duration and severity at each follow-up visit (based on scale of mild, moderate and severe) in those eyes which develop SEIs
Degree of Bulbar conjunctival Injection | 21 days
  Degree of bulbar conjunctival injection (redness of the eye) (as determined by the Efron scale) at each follow-up visit
Second eye involvment | 14 days
  Second eye involvement - incidence for the study duration and severity at each visit up to Day 14(measured as degree of bulbar injection using Efron scale) in the baseline culture negative fellow eyes, which turned culture positive during the study up to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Jay S Pepose, MD, PhD, Study Director — Lifelong Vision Foundation; Parag A Majmudar, MD, Principal Investigator — Chicago Cornea Consultants; Kevin L Waltz, OD, MD, Principal Investigator — Eye Surgeons of Indiana; Jai Parekh, MD, MBA, Principal Investigator — Brar-Parekh Eye Associates; Mujtaba A Qazi, MD, Principal Investigator — Lifelong Vision Foundation; John Sheppard, MD, Principal Investigator — Virginia Eye Consultants; Ruben L BonSiong, MD, Principal Investigator — Philippines General Hospital
Locations (1):
- Lifelong Vision Foundation, Chesterfield, Missouri, United States